CLINICAL TRIAL: NCT04171726
Title: Rotterdam EDOXaban Leaflet Evaluation in Patients After Transcatheter Aortic Valve Implantation
Acronym: REDOX-TAVI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Principal investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDOX TAVI
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Stenosis
Keywords: Thrombosis; Aortic Valve Stenosis; Heart Valve Diseases; Ventricular Outflow Obstruction; Cardiovascular Diseases; Embolism and Thrombosis; Vascular Diseases; Heart Diseases; Factor Xa Inhibitors; Anticoagulants
MeSH Terms: conditions — Aortic Valve Stenosis; Thrombosis; Heart Valve Diseases; Ventricular Outflow Obstruction; Cardiovascular Diseases; Embolism and Thrombosis; Vascular Diseases; Heart Diseases | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Edoxaban (Experimental): treatment with edoxaban
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — A non-vitamin K antagonist (VKA) oral anticoagulant that selectively inhibits factor Xa.

SUMMARY:
A single-center, investigator-initiated, single arm interventional study in patients undergoing transfemoral transcatheter aortic valve replacement (TAVR) in the Erasmus Medical Center in Rotterdam (NL). Study population will be patients undergoing TAVR with no formal indication for oral anticoagulant (OAC) and no dual antiplatelet therapy (DAPT) requirement for coronary stents. Primary endpoint is the incidence of leaflet thickening on MSCT after three months of edoxaban treatment.

DETAILED DESCRIPTION:
Rationale: Thromboembolic- and bleeding events can occur after TAVI and can have great consequences. There is currently no evidence-based guideline on prevention of thromboembolic events after TAVI and the current standard of care with DAPT 3-6 months is based on expert opinion. Recently multislice computed tomography (MSCT) studies identified bioprosthesis leaflet thickening and impaired leaflet motion after TAVI. The goal of this study is to investigate whether in TAVI patients, treatment with edoxaban leads to a reduction in leaflet thickening incidence after 3 months and whether it is safe and clinically efficient.

Objective: To investigate whether treatment with edoxaban leads to a decrease in incidence of leaflet thickening and is clinical efficient and safe.

Study design: A single-center, investigator-initiated, open-label, observational study.

Study population: Patients undergoing transfemoral transcatheter aortic valve replacement in the Erasmus University Medical Center with no formal novel oral anticoagulants/vitamin-K-antagonist (NOAC/VKA) indication.

Intervention (if applicable): Patients will be treated with edoxaban for a period of 3 months following TAVI. Afterwards they will switch to acetylsalicylic acid.

Main study parameters/endpoints: The incidence of leaflet thickening on MSCT 3 months after TAVI and edoxaban treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Thus far edoxaban has proven to be safe and non-inferior to treatment with warfarin in several indications. The role of anticoagulant agents in TAVI still has to be unravelled. Subjects participating in this trial are possibly at higher risk for bleeding complications than patients being treated with dual antiplatelet therapy after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Completed successful elective TAVI for severe native aortic valve stenosis with any commercially-available transcatheter heart valve (THV).

  * Correct positioning of a single prosthetic heart valve
  * Device success, defined by:

    * Mean aortic valve gradient < 20 mmHg
    * Peak transvalvular velocity < 3.0 m/s
    * Aortic valve regurgitation of 2 or less
* No periprocedural complications.

  * No overt stroke
  * No uncontrolled bleeding
  * No major vascular complication defined by the Valve academic research committee 2 (VARC-2) consensus
* No formal indication for oral anticoagulation

  * Prevention of thromboembolic complications in patients with atrial fibrillation
  * Prevention for recurrent venous thromboembolism
  * Prevention for recurrent pulmonary embolism

Exclusion Criteria:

* History of life-threatening or major bleeding event ≥ Bleeding academic research committee (BARC) 3b definitions within the last year.
* Conditions with a high risk of bleeding

  * Active peptic ulcer or upper gastrointestinal bleeding (< 3 months)
  * Malignancy with high risk of bleeding
  * Recent unresolved brain of spinal injury
  * Spinal or ophthalmic surgery within last 3 months prior to enrolment
  * Intracranial haemorrhage
  * Esophagal varices
  * Arteriovenous malformations with high risk of bleeding
  * Vascular aneurysms
  * Major intraspinal or intracerebral vascular abnormalities
* Hypersensitivity or contraindications to edoxaban
* No percutaneous coronary intervention within 6 months prior to randomization (requiring DAPT after TAVR)
* Dialysis-dependency or glomerular filtration rate < 30 mL/min at time of enrollment
* Active bleeding or bleeding diathesis including thrombocytopenia (platelet count < 50.000 cells/UL), thromboasthenia, haemophilia or von Willebrand disease
* Patients unable to adhere to or complete the investigational protocol for any reason including but not limited to geographical residence, psychiatric condition or life-threatening disease
* Pregnant or breast-feeding subjects
* Current participation in clinical trials that potentially interfere with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of aortic valve leaflet thickening after TAVI as assessed by cardiac 4D computed tomography scan (4DCT) | 3 months after TAVI
  total of participants with aortic valve thickening after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Van Mieghem, MD, PhD, Principal Investigator — Erasmusm MC
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Background] Sondergaard L, De Backer O, Kofoed KF, Jilaihawi H, Fuchs A, Chakravarty T, Kashif M, Kazuno Y, Kawamori H, Maeno Y, Bieliauskas G, Guo H, Stone GW, Makkar R. Natural history of subclinical leaflet thrombosis affecting motion in bioprosthetic aortic valves. Eur Heart J. 2017 Jul 21;38(28):2201-2207. doi: 10.1093/eurheartj/ehx369. PMID 28838044
- [Background] Chakravarty T, Sondergaard L, Friedman J, De Backer O, Berman D, Kofoed KF, Jilaihawi H, Shiota T, Abramowitz Y, Jorgensen TH, Rami T, Israr S, Fontana G, de Knegt M, Fuchs A, Lyden P, Trento A, Bhatt DL, Leon MB, Makkar RR; RESOLVE; SAVORY Investigators. Subclinical leaflet thrombosis in surgical and transcatheter bioprosthetic aortic valves: an observational study. Lancet. 2017 Jun 17;389(10087):2383-2392. doi: 10.1016/S0140-6736(17)30757-2. Epub 2017 Mar 19. PMID 28330690
- [Derived] Adrichem R, van Wiechen MP, Knol WG, Hokken TW, Ooms JF, van den Dorpel MMP, Verhemel S, Kardys I, Nuis RJ, Daemen J, Hirsch A, Budde RPJ, Van Mieghem NM. Edoxaban Monotherapy and Incidence of Transcatheter Heart Valve Leaflet Thrombosis - The Rotterdam Edoxaban (REDOX) Study. Catheter Cardiovasc Interv. 2025 Feb;105(2):375-384. doi: 10.1002/ccd.31300. Epub 2024 Nov 22. PMID 39575924
- [Derived] van Wiechen MP, El Azzouzi I, Knol WG, Adrichem R, Hokken TW, Ooms JF, de Ronde-Tillmans MJ, Daemen J, de Jaegere PP, Hirsch A, Budde RPJ, Van Mieghem NM. Leaflet Thickening and Motion After Transcatheter Aortic Valve Replacement: Design and Rationale of the Rotterdam Edoxaban Trial. Cardiovasc Revasc Med. 2022 Nov;44:67-70. doi: 10.1016/j.carrev.2022.06.011. Epub 2022 Jun 17. PMID 35787831